CLINICAL TRIAL: NCT03533569
Title: Early Biomarkers for ARthritic PAIN to Guide Improved Treatments for Arthritis (ARPAIN) Study
Brief Title: Early Biomarkers for ARthritic PAIN to Guide Improved Treatments for Arthritis
Acronym: ARPAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Wellcome Trust (Other); Rosetrees Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17.0192; 17/LO/1894 (Other: Integrated Research Application System (UK))
Record Dates: First submitted 2018-04-17; First posted 2018-05-23 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Knee; Rheumatoid Arthritis; Spondyloarthritis; Psoriatic Arthritis
Keywords: pain; inflammation
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic; Pain; Inflammation | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for protein and DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Osteoarthritis: Participants with an established diagnosis of knee osteoarthritis
  Interventions: Procedure: Intra-articular corticosteroid injection
- Rheumatoid arthritis: Participants with an established diagnosis of rheumatoid arthritis
  Interventions: Procedure: Intra-articular corticosteroid injection
- Spondyloarthritis or psoriatic arthritis: Participants with an established diagnosis of spondyloarthritis or psoriatic arthritis
  Interventions: Procedure: Intra-articular corticosteroid injection
- Case controls: Participants with no arthritis or knee pain as controls

INTERVENTIONS:
Procedure: Intra-articular corticosteroid injection — Participants with arthritis will undergo usual care with knee synovial fluid aspiration followed by intra-articular corticosteroid injection
  Groups: Osteoarthritis; Rheumatoid arthritis; Spondyloarthritis or psoriatic arthritis

SUMMARY:
Osteoarthritis (OA) is a condition affecting the whole joint and is a major cause of pain and disability worldwide. Although OA is very common, the initial steps which lead to the development of pain and tissue damage are not fully understood. In this study participants will be investigated for markers in the blood, joint and urine in people who have a diagnosis of osteoarthritis or inflammatory arthritis and are receiving a steroid injection for their condition. Markers will be evaluated in participants with osteoarthritis compared with other types of arthritis, including rheumatoid arthritis and spondyloarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis worldwide. OA causes major disability and pain and places a huge financial burden on healthcare worldwide. In recent work, the gene expression profile of bone marrow lesions (BML) in osteoarthritis has been evaluated. BML in OA have a novel gene expression profile which includes genes involved in inflammation, neurogenesis and matrix turnover. The plan is to investigate the functional significance of the genes found at the protein biomarker level in studies of joint tissue, blood and urine from participants with knee OA and compare these changes with participants who have other forms of arthritis, including rheumatoid arthritis and spondyloarthritis.

A study amendment was added in April 2020 due to Covid-19. We are studying up to 150 additional participants with or without inflammatory conditions who are being treated with immunomodulatory drugs compared with participants who are not on immunomodulators. We will be evaluating the course of Covid-19 infection in people without autoimmune inflammatory conditions, compared with people who have autoimmune inflammatory diseases who are on immunomodulators.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for OA patients:

* Fulfilling the American College of Rheumatology (ACR) criteria for the diagnosis of knee osteoarthritis
* Symptomatic knee pain
* On usual care for knee osteoarthritis including paracetamol and/or NSAIDs

Inclusion criteria for Inflammatory Arthritis Patients:

* Fulfilling the American College of Rheumatology (ACR) criteria for the diagnosis of inflammatory arthritis i.e. rheumatoid arthritis (Anti-CCP antibodies & Rheumatoid Factor checked ), psoriatic arthritis or spondyloarthropathy
* Symptomatic knee pain
* On usual care for arthritis including disease-modifying anti-rheumatic drugs (DMARDs), paracetamol and/or NSAIDs

Exclusion Criteria:

* Other rheumatological diagnosis e.g. systemic lupus erythematosus, fibromyalgia, Polymyalgia Rheumatica, Gout, Giant Cell Arteritis, Sjogren's syndrome
* History of uncontrolled depression
* Recent surgery
* Uncontrolled ischaemic heart disease
* Uncontrolled diabetes mellitus
* Alcohol consumption > 14 units/week as per UK National guidelines
* Participants unable to give full informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes participants with an established diagnosis of knee osteoarthritis, rheumatoid arthritis, spondyloarthritis or psoriatic arthritis. A control group without arthritis or knee pain serves as the comparator group
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-04-02 (Estimated); Study Completion 2022-04-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Numerical Rating Scale (NRS) for pain in target knee after 3 months | Baseline (Visit 1) and 3 months after treatment (Visit 2)
  Pain outcome measure. The Numerical Rating Scale for pain has a range of 0 - 10, with the lowest score being 0 and the highest rating at 10.The pain rating will be reported by the participants for their symptomatic knee

SECONDARY OUTCOMES:
Change in Biomarkers 3 months following treatment | Baseline (Visit 1) and 3 months after treatment (Visit 2)
  Protein measurements in serum, urine and synovial fluid for type II collagen degradation products in the samples. The levels of type II collagen degradation products may range from 0 to greater than 500 ng/mmol, depending on the stage and severity of the condition

CONTACTS AND LOCATIONS:
Overall Officials: Nidhi Dr Sofat, MD, PhD, Principal Investigator — St George's, University of London
Locations (1):
- St George's Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
All data will be published and open access after completion of the study.